CLINICAL TRIAL: NCT02587910
Title: Melanole, a Nigella Sativa (Black Seed) Extract for the Treatment of Gastroesophageal Reflux Disease
Brief Title: Melanole, a Dietary Supplement, for the Treatment of Gastroesophageal Reflux Disease
Acronym: GERDMeDS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lebanese American University (Other)
Responsible Party: Principal Investigator, Dr Rajaa Chatila, Associate Professor of Medicine, Lebanese American University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LAUMCRH.RC3.23/Sep/2015
Record Dates: First submitted 2015-10-17; First posted 2015-10-27 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Nigella sativa oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-invasive arm (Placebo Comparator): Participants in this arm, who fit the inclusion criteria and have a GERD Q score of 3 or more, will be randomized to receive either Melanole, a herbal derived melanin, 300 mg, 2 capsules three times a day or placebo for 10 days.To assess the symptomatic improvement, GERD Q score will be calculated on day 0 (before administration of the product) and then on days 11 and 30 having taken the product for 10 days.
  Interventions: Dietary Supplement: Melanole for GERD treatment; Dietary Supplement: Placebo
- Invasive arm (Placebo Comparator): Participants in this arm will undergo a 24-hour pH monitoring before administration of Melanole, the herbal melanin or placebo. They will then be randomized to receive either Melanole or placebo for 10 days. pH metry will be repeated between days 7 and 10 from the study product or placebo.
  Interventions: Dietary Supplement: Melanole for GERD treatment; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Melanole for GERD treatment — Melanole is given orally as 2 capsules TID 5 minutes before each meal
  Other Names: GERDMeDS; Melanole; Nigella sativa
Dietary Supplement: Placebo — Placebo is given orally as 2 capsules TID 5 minutes before each meal

SUMMARY:
Melanole, a Nigella sativa (Black Seed) extract , is studied for the treatment of GERD. Participants, who meet the inclusion criteria, will be divided into two arms.

Arm 1: Subjects who meet criteria for GERD will undergo 24 hour pH monitoring.

Arm 2: Subjects who meet criteria for GERD and who undergo only symptomatic monitoring of GERD on treatment.

All participants will be evaluated before and after the administration of the study product.

DETAILED DESCRIPTION:
Volunteers were recruited in Lebanese American University campuses. Those who fit the inclusion criteria were allowed to choose between two arms: invasive or non-invasive procedures.

Volunteers who chose to enroll in the non-invasive arm were given the study product directly after completing the GERD Q questionnaire. A follow-up by phone was done on day 0, 3 , 6 and 11. GERD Q questionnaire was repeated on days 11 and 28 along with a satisfaction rating. Adverse events were reported on a log sheet.

Concerning the invasive arm, volunteers were given an appointment at Lebanese American University Medical Center Rizk Hospital to place the 24h pH-metry, after study product was administered. After 7-10 days, the 24h pH monitoring was done again.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with age (18-60) with GerdQ score ≥3

Exclusion Criteria:

* Patients younger than 18 year or older than 60years
* Dysphagia, odynophagia, weight loss, palpable mass
* Nonsteroidal antiinflammatory drug intake (including aspirin)
* History of hyperparathyroidism
* Coronary artery disease or congestive heart failure
* History of liver disease
* History of renal disease
* Pregnancy
* History of active cancer or chemotherapy
* History of intake of any drug known to affect reflux (phenothiazine, anticholinergic, nitrates, calcium channel blockers and proton pump inhibitors) within 14 days of inclusion to the study
* Prior esophageal or gastric surgeries of any type
* Allergy to black seeds or Lidocaine
* Any important nasal anatomical anomaly
* Any use of chronic medications for chronic medical conditions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-04 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Change of GERD Q scores from baseline at day 11 as measured by the GERD Q questionnaire | GERD Q questionnaire and score were measured at day 0, then remeasured on day 11
  GERD Q scores on day 0 and day 11 were compared and the difference was analyzed

SECONDARY OUTCOMES:
Number of patients experiencing a reduction in the number of reflux episodes by 10 or more where the reflux episode is defined as a pH reading less than 4, as well was a reduction in the total time where the pH in esophagus is less than 4. | The pH metry study was conducted at day 0 ,and then reconducted on day 11
  Number of reflux episodes and total number of time where the pH in esophagus was less than 4 were calculated on days 0 and 11, and then analyzed to check how the given treatment affects the results
Number of participants with treatment-related adverse events as reported during follow-up on days 3, 6 and 11. | Adverse events were recorded on days 3, 6 and 11

CONTACTS AND LOCATIONS:
Overall Officials: Rajaa Chatila, MD, Principal Investigator — Lebanese American University; Hani Dimassi, PhD, Principal Investigator — Lebanese American University; Mohamad Mroueh, PhD, Principal Investigator — Lebanese American University
Locations (2):
- Lebanon (2):
  - Lebanese American University, Beirut
  - Lebanese American University, Byblos

REFERENCES:
- [Background] Spiegel B. Diagnostic testing in extraesophageal GERD: another case of "furor medicus"? Am J Gastroenterol. 2013 Jun;108(6):912-4. doi: 10.1038/ajg.2013.80. PMID 23735914
- [Background] Magdy MA, Hanan el-A, Nabila el-M. Thymoquinone: Novel gastroprotective mechanisms. Eur J Pharmacol. 2012 Dec 15;697(1-3):126-31. doi: 10.1016/j.ejphar.2012.09.042. Epub 2012 Oct 7. PMID 23051678
- [Background] Dent J, El-Serag HB, Wallander MA, Johansson S. Epidemiology of gastro-oesophageal reflux disease: a systematic review. Gut. 2005 May;54(5):710-7. doi: 10.1136/gut.2004.051821. PMID 15831922
- [Background] Jones R, Junghard O, Dent J, Vakil N, Halling K, Wernersson B, Lind T. Development of the GerdQ, a tool for the diagnosis and management of gastro-oesophageal reflux disease in primary care. Aliment Pharmacol Ther. 2009 Nov 15;30(10):1030-8. doi: 10.1111/j.1365-2036.2009.04142.x. Epub 2009 Sep 8. PMID 19737151
- [Background] Ahmad A, Husain A, Mujeeb M, Khan SA, Najmi AK, Siddique NA, Damanhouri ZA, Anwar F. A review on therapeutic potential of Nigella sativa: A miracle herb. Asian Pac J Trop Biomed. 2013 May;3(5):337-52. doi: 10.1016/S2221-1691(13)60075-1. PMID 23646296
- [Background] Al Mofleh IA, Alhaider AA, Mossa JS, Al-Sohaibani MO, Al-Yahya MA, Rafatullah S, Shaik SA. Gastroprotective effect of an aqueous suspension of black cumin Nigella sativa on necrotizing agents-induced gastric injury in experimental animals. Saudi J Gastroenterol. 2008 Jul;14(3):128-34. doi: 10.4103/1319-3767.41731. PMID 19568521